CLINICAL TRIAL: NCT01452568
Title: Early Anticoagulation Therapy After Bioprosthetic Aortic Valve Implantation: Comparing Warfarin Versus Aspirin
Brief Title: Anticoagulant After Implantation of Biological Aortic Valve Comparing With Aspirin
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Nikolaj B. Lilleoer, Clinical Project Coordinator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01-080/04; (KF) 01-080/04 (Other: Science Ethics Committee Copenhagen)
Record Dates: First submitted 2009-09-22; First posted 2011-10-17 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Thromboembolism; Bleeding
Keywords: Thromboembolic complications; Bleeding complications; Haemorrhagic complications; Anticoagulant therapy; Aspirin; biological Aorta Valve
MeSH Terms: conditions — Thromboembolism; Hemorrhage | interventions — Aspirin; aspirin, magnesium oxide combination; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aspirin (Experimental): Aspirin 150mg daily, starting day 1 after surgery, for three months.
  Interventions: Drug: Aspirin
- Warfarin (Active Comparator): Warfarin daily dosage to International normalized ratio(INR) value between 2,0 to 3,0.
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Aspirin — 150mg/daily for three months, starting day after surgery
  Other Names: Magnyl, Acetyl salicylic acid
  Arms: Aspirin
Drug: Warfarin — Warfarin daily dosage to obtain an INR in between 2,0 to 3,0. Started the day after surgery and continued for three months.
  Other Names: marevan
  Arms: Warfarin

SUMMARY:
The optimal medical strategy for prevention of thromboembolic events after bioprosthetic aorta valve replacement (BAVR) remains controversial.

The aim of this trial was to compare warfarin therapy (target INR of 2.0 to 3.0) against aspirin 150mg daily as antithrombotic therapy for the first three months after BAVR with or without concomitant coronary artery bypass grafting (CABG). The aim was to evaluate thromboembolic complications, bleeding complications and death.

ELIGIBILITY:
Inclusion criteria:

* Patients with aortic valve disease where there is indication for implantation of a biological stented aortic valve with or without coronary bypass surgery.
* Age 60 years Sinus rhythm

Exclusion Criteria:

* Patients planned for double valve surgery
* Patients with active endocarditis
* Patients with atrial fibrillation/flutter
* Patients in anticoagulation treatment of other reason.
* Patients with previous cerebrovascular accidents or insults.
* Patients with TCI
* Patients with hypercoagulable conditions, disseminated intervascular coagulation, haemophilia or any other blood coagulapathy or related condition, whereby the blood coagulation process is not readily controllable
* Patients with pacemaker
* Any other disease than valve disease that will considerably increase the operative risk and increase the probability that the patient dies within one year after the operation, for example because of terminal cancer
* Patients that is HIV-positive or have active AIDS
* Patients that are known drug abuser
* Patients in chronic haemodialysis or other types of dialysis

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2005-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Haemorrhagic complications | 3 months
  Bleeding complications
Thromboembolic complications | 3 months
  TCI, stroke, Myocardial infarction (MI), Pulmonary embolism, Deep vein thrombosis (DVT) , peripheral arterial embolism, intra-cardiac thrombus formation. We expected statistically fewer thromboembolic events in the groups receiving anticoagulation with warfarin than the aspirin only groups.

SECONDARY OUTCOMES:
Echocardiographic findings before surgery, before discharge and 3 months after implantation | 3 months
Registration of surgical data and postoperative complications | 3 months
All cause mortality | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter S Olsen, MD, DMSc, Principal Investigator — Cardiothoracic Surgery, Rigshospitalet, University of Copenhagen; Nikolaj B Lilleør, Principal Investigator — Cardiothoracic Surgery, Rigshospitalet, University of Copenhagen; Sulman Rafiq, Study Chair — Cardiothoracic Surgery, Rigshospitalet, University of Copenhagen